CLINICAL TRIAL: NCT05701163
Title: Assessing the Effect of Abstinence Period on Semen Parameters
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There is no funds available for the study.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-10024093
Record Dates: First submitted 2022-12-23; First posted 2023-01-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Healthy males with no significant comorbidities, aged 20-45 years who are able to produce a semen sample by masturbation.
  Interventions: Other: Abstinence followed by semen sample collection.

INTERVENTIONS:
Other: Abstinence followed by semen sample collection. — Abstinence is the intervention. Semen samples will be collected after abstinence periods.

SUMMARY:
The goal of this study is to learn about the impact of abstinence periods on sperm quality in healthy males 20-45 years of age with no significant comorbidities who are able to produce a semen sample via masturbation. The main question it aims to answer is:

• Do shorter abstinence periods result in improved semen quality?

Participants will provide semen samples for analysis following abstinence periods of 7 days, 5 days, 2 days, 1 day, and 3 hours.

DETAILED DESCRIPTION:
Participant Duration: Total length of time on study per subject is 14 days (including 5 days of visit required for sample production). Subjects do not need to complete the visits in order but need to document abstinence period prior to sample production. No follow up will be needed after the study.

Primary Objective: The primary objective is to examine the differences in semen analysis parameters after varying abstinence periods (7 days, 5 days, 2 days, 1 day, 3 hours).

Secondary Objectives: The secondary objective(s) is to assess changes in sperm DNA fragmentation after varying abstinence periods (7 days, 5 days, 2 days, 1 day, 3 hours).

ELIGIBILITY:
Inclusion Criteria:

* Males, aged 20-45 years
* Healthy, no significant comorbidities
* Able to produce a semen sample by masturbation
* Total sperm count ≥ 1 million sperm
* Abnormal sperm DNA fragmentation (TUNEL assay value ≥ 20%)

Exclusion Criteria:

* Age < 20 or > 45 years
* Significant comorbidities, including significant cardiac, pulmonary, gastrointestinal, hematologic, or neurologic disease
* Total sperm count < 1 million sperm
* Aspermia (semen volume = 0)
* Normal sperm DNA fragmentation (TUNEL assay value < 20%)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 0 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2028-02-05 (Estimated); Study Completion 2028-02-05 (Estimated)

PRIMARY OUTCOMES:
Change in semen analysis parameters based on different abstinence periods: volume | 7 days, 5 days, 2 days, 1 day, 3 hours
  The primary objective is to examine the differences in semen analysis parameters (volume in mL) after varying abstinence periods (7 days, 5 days, 2 days, 1 day, 3 hours).
Change in semen analysis parameters based on different abstinence periods: sperm concentration | 7 days, 5 days, 2 days, 1 day, 3 hours
  The primary objective is to examine the differences in semen analysis parameters (sperm concentration measured in million sperm/mL) after varying abstinence periods (7 days, 5 days, 2 days, 1 day, 3 hours).
Change in semen analysis parameters based on different abstinence periods: motility | 7 days, 5 days, 2 days, 1 day, 3 hours
  The primary objective is to examine the differences in semen analysis parameters (motility measured as a percentage) after varying abstinence periods (7 days, 5 days, 2 days, 1 day, 3 hours).

SECONDARY OUTCOMES:
Change in sperm DNA fragmentation based on different abstinence periods | 7 days, 5 days, 2 days, 1 day, 3 hours
  The secondary objective(s) is to assess changes in sperm DNA fragmentation after varying abstinence periods (7 days, 5 days, 2 days, 1 day, 3 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No